CLINICAL TRIAL: NCT00787839
Title: Screening for Prediabetes and Early Diabetes in Primary Care
Brief Title: Opportunistic Screening for Prediabetes and Early Diabetes in Primary Care
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 07-138
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes Mellitus; Prediabetic State
Keywords: type 2 diabetes mellitus; prediabetic state; mass screening; glucose tolerance test
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Atlanta VA Medical Center patients who meet criteria for screening for prediabetes and early diabetes based on standard guidelines of the VA, the American Diabetes Association, and the National Institutes of Health
  Interventions: Other: Glucose challenge test; Other: Glucose tolerance test

INTERVENTIONS:
Other: Glucose challenge test — At a first outpatient visit, at different times of the day and without a prior fast, subjects will have a 50 gram glucose drink followed by measurement of plasma and capillary glucose along with A1c one hour later. They will also fill out questionnaires. At a second outpatient visit, in the morning after fasting overnight, they will have a 75 gram oral glucose tolerance test.
Other: Glucose tolerance test — Subjects found to have diabetes or prediabetes on the initial glucose tolerance test may be requested to have a repeat glucose tolerance test and A1c.

SUMMARY:
People who might have prediabetes or unrecognized diabetes will be screened for these problems at an outpatient visit. For screening, they will take a sugary drink containing 50 grams of glucose, and have a blood sample one hour later. The blood sample will be tested for glucose and A1c (a measure of blood glucose over the previous two months). They will also fill out questionnaires that ask about their health history and how they would feel about exercising and trying to lose weight if they are found to have prediabetes or diabetes. At a subsequent visit, they will have an oral glucose tolerance test (OGTT) - a blood sample, then a sugary drink containing 75 grams of glucose, and a repeat blood sample 2 hours later. We will evaluate the costs of finding out if people have prediabetes or diabetes. For people who are found to have these problems, we will also evaluate how well their doctors treat these problems.

DETAILED DESCRIPTION:
RELEVANCE TO VETERANS' HEALTH: Lack of a good strategy to identify prediabetes - probably ~10 years prior to the development of diabetes that is recognized clinically - may be the greatest present impediment to diabetes care. We are developing a new way to screen for prediabetes, and it should constitute a major opportunity to improve the health of ~4 million veterans; early recognition of glucose intolerance would permit institution of preventive strategies which are efficacious, convenient, and cost-effective - improving the health of individual veterans, reducing diabetes-related health care resource use and costs for the VA, and helping to spare VA funds for management of other disorders.

BACKGROUND: Prediabetes is a major public health problem which confers risk of diabetes and cardiovascular disease (CVD), but veterans with prediabetes are not detected, and cannot receive interventions to reduce their risks; CVD events, health resource use, and cost all rise before diabetes is diagnosed. Diabetes can be prevented or delayed by lifestyle change or medication, but since we do not identify prediabetes, glucose intolerance progresses for 5-10 years, and many patients have early diabetes complications and increased CVD risk when they are finally recognized. We are developing a new screening test for prediabetes, a "glucose challenge test" (GCT): patients have a 50g oral glucose challenge at any time of day, regardless of meal status, with a single 1 hr sample. If the GCT exceeds a cutoff, they have a 75g oral glucose tolerance test after an overnight fast, with 0 and 2 hr samples (OGTT). Our GCRC-based Preliminary Data show ROC AUC 0.83 (70% specificity, 82% sensitivity) and $51 per case identified; the GCT should constitute an effective, convenient, inexpensive, cost-effective screen for prediabetes - a critical indicator of individual, VA health care system, and societal risk.

OBJECTIVES: To translate our findings into improved health for VA patients, the GCT will need to be implemented in VA primary care settings - where practitioners often do not screen for prediabetes, or manage diabetes optimally. Such barriers must be overcome in order to conduct definitive studies aimed to show that use of the GCT to detect prediabetes (and previously unrecognized diabetes) in primary care leads to improved outcomes. Thus, VA policies for system-wide implementation of GCT screening must be preceded by logical next steps: validation and demonstration of likely cost-effectiveness.

METHODS: AIM #1. Validation: (A) To establish feasibility, we will interact with VA primary care providers to solve logistical problems, and determine optimal screening strategies. (B) To assess test performance, we will (a) perform GCTs and measure A1c in ~1,800 patients, (b) evaluate OGTTs in all subjects, and (c) compare sensitivity, specificity, and ROC curves from GCT vs. A1c or "predictive model" screening in primary care to those in our GCRC studies. Availability of this dataset will also permit (d) subsequent management of diabetes/prediabetes to be evaluated relative to standardized guidelines. AIM #2. Costs: To evaluate impact, we will (a) capture the costs of diagnostic tests, staff effort, and patient time; (b) express cost per case identified from both VA health system and societal perspectives; and (c) compare GCT vs. alternative strategies with a wide range of assumptions about false-(+)/false-(-) costs to reflect downstream cost implications of test imperfections. Engagement with this process will also provide (d) for those study patients with prediabetes who go on to develop diabetes, an opportunity to explore VA resource use and costs before and after the diagnosis of diabetes. This will provide preliminary data for subsequent proposals to compare resource use and costs vs. those of other VA patients who are newly diagnosed with diabetes in settings where there is no screening for prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* veteran status,
* ambulatory outpatient at Atlanta VA Medical Center,
* visit to primary care clinic, AND
* meet criteria for screening (age >= 45 years or other risk factors [body mass index >=25 or hypertension or systolic blood pressure >=140 or HDL cholesterol <35 in men or <45 in women or fasting triglycerides >250 or first-degree relative with diabetes or minority race or minority ethnicity or history of diabetes during pregnancy or history of having a baby weighing >9 pounds or history of polycystic ovary syndrome])

Exclusion Criteria:

* known to have diabetes, OR
* taking steroids OR pregnant, OR
* not well enough to have worked during the previous week (actual employment not necessary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: initial primary study population will be drawn primarily from veterans receiving primary care at the Decatur Clinic CBOC in metropolitan Atlanta, GA
Sampling Method: Non-Probability Sample
Enrollment: 1939 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S Phillips, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

REFERENCES:
- [Result] Twombly JG, Long Q, Zhu M, Wilson PW, Narayan KM, Fraser LA, Webber BC, Phillips LS. Diabetes care in black and white veterans in the southeastern U.S. Diabetes Care. 2010 May;33(5):958-63. doi: 10.2337/dc09-1556. Epub 2010 Jan 26. PMID 20103548
- [Result] Ziemer DC, Kolm P, Weintraub WS, Vaccarino V, Rhee MK, Twombly JG, Narayan KM, Koch DD, Phillips LS. Glucose-independent, black-white differences in hemoglobin A1c levels: a cross-sectional analysis of 2 studies. Ann Intern Med. 2010 Jun 15;152(12):770-7. doi: 10.7326/0003-4819-152-12-201006150-00004. PMID 20547905
- [Result] Rhee MK, Herrick K, Ziemer DC, Vaccarino V, Weintraub WS, Narayan KM, Kolm P, Twombly JG, Phillips LS. Many Americans have pre-diabetes and should be considered for metformin therapy. Diabetes Care. 2010 Jan;33(1):49-54. doi: 10.2337/dc09-0341. Epub 2009 Oct 6. PMID 19808929
- [Result] Olson DE, Rhee MK, Herrick K, Ziemer DC, Twombly JG, Phillips LS. Screening for diabetes and pre-diabetes with proposed A1C-based diagnostic criteria. Diabetes Care. 2010 Oct;33(10):2184-9. doi: 10.2337/dc10-0433. Epub 2010 Jul 16. PMID 20639452
- [Result] Fraser LA, Twombly J, Zhu M, Long Q, Hanfelt JJ, Narayan KM, Wilson PW, Phillips LS. Delay in diagnosis of diabetes is not the patient's fault. Diabetes Care. 2010 Jan;33(1):e10. doi: 10.2337/dc09-1129. No abstract available. PMID 20040660
- [Result] Lin E, Liang Z, Frediani J, Davis SS Jr, Sweeney JF, Ziegler TR, Phillips LS, Gletsu-Miller N. Improvement in ss-cell function in patients with normal and hyperglycemia following Roux-en-Y gastric bypass surgery. Am J Physiol Endocrinol Metab. 2010 Nov;299(5):E706-12. doi: 10.1152/ajpendo.00405.2010. Epub 2010 Aug 17. PMID 20716694
- [Result] Chatterjee R, Narayan KM, Lipscomb J, Phillips LS. Screening adults for pre-diabetes and diabetes may be cost-saving. Diabetes Care. 2010 Jul;33(7):1484-90. doi: 10.2337/dc10-0054. PMID 20587721
- [Result] Twombly JG, Long Q, Zhu M, Fraser LA, Olson DE, Wilson PW, Narayan KM, Phillips LS. Validity of the primary care diagnosis of diabetes in veterans in the southeastern United States. Diabetes Res Clin Pract. 2011 Mar;91(3):395-400. doi: 10.1016/j.diabres.2010.11.001. Epub 2010 Nov 26. PMID 21112654
- [Result] Phillips LS, Ziemer DC, Kolm P, Weintraub WS, Vaccarino V, Rhee MK, Chatterjee R, Narayan KM, Koch DD. Glucose challenge test screening for prediabetes and undiagnosed diabetes. Diabetologia. 2009 Sep;52(9):1798-807. doi: 10.1007/s00125-009-1407-7. Epub 2009 Jun 26. PMID 19557386
- [Result] Shikany JM, Tinker LF, Neuhouser ML, Ma Y, Patterson RE, Phillips LS, Liu S, Redden DT. Association of glycemic load with cardiovascular disease risk factors: the Women's Health Initiative Observational Study. Nutrition. 2010 Jun;26(6):641-7. doi: 10.1016/j.nut.2009.08.014. Epub 2010 Jan 6. PMID 20053533
- [Result] Buse JB. Screening for diabetes and prediabetes with proposed A1C-based diagnostic criteria: comment on Olson et al. Diabetes Care. 2010 Dec;33(12):e174; author reply e175. doi: 10.2337/dc10-1720. No abstract available. PMID 21115761
- [Result] Margolis KL, Wei F, de Boer IH, Howard BV, Liu S, Manson JE, Mossavar-Rahmani Y, Phillips LS, Shikany JM, Tinker LF; Women's Health Initiative Investigators. A diet high in low-fat dairy products lowers diabetes risk in postmenopausal women. J Nutr. 2011 Nov;141(11):1969-74. doi: 10.3945/jn.111.143339. Epub 2011 Sep 21. PMID 21940514
- [Result] Tinker LF, Sarto GE, Howard BV, Huang Y, Neuhouser ML, Mossavar-Rahmani Y, Beasley JM, Margolis KL, Eaton CB, Phillips LS, Prentice RL. Biomarker-calibrated dietary energy and protein intake associations with diabetes risk among postmenopausal women from the Women's Health Initiative. Am J Clin Nutr. 2011 Dec;94(6):1600-6. doi: 10.3945/ajcn.111.018648. Epub 2011 Nov 9. PMID 22071707
- [Result] Chlebowski RT, McTiernan A, Wactawski-Wende J, Manson JE, Aragaki AK, Rohan T, Ipp E, Kaklamani VG, Vitolins M, Wallace R, Gunter M, Phillips LS, Strickler H, Margolis K, Euhus DM. Diabetes, metformin, and breast cancer in postmenopausal women. J Clin Oncol. 2012 Aug 10;30(23):2844-52. doi: 10.1200/JCO.2011.39.7505. Epub 2012 Jun 11. PMID 22689798
- [Result] Ma Y, Hebert JR, Manson JE, Balasubramanian R, Liu S, Lamonte MJ, Bird CE, Ockene JK, Qiao Y, Olendzki B, Schneider KL, Rosal MC, Sepavich DM, Wactawski-Wende J, Stefanick ML, Phillips LS, Ockene IS, Kaplan RC, Sarto GE, Garcia L, Howard BV. Determinants of racial/ethnic disparities in incidence of diabetes in postmenopausal women in the U.S.: The Women's Health Initiative 1993-2009. Diabetes Care. 2012 Nov;35(11):2226-34. doi: 10.2337/dc12-0412. Epub 2012 Jul 25. PMID 22833490
- [Result] You NC, Chen BH, Song Y, Lu X, Chen Y, Manson JE, Kang M, Howard BV, Margolis KL, Curb JD, Phillips LS, Stefanick ML, Tinker LF, Liu S. A prospective study of leukocyte telomere length and risk of type 2 diabetes in postmenopausal women. Diabetes. 2012 Nov;61(11):2998-3004. doi: 10.2337/db12-0241. Epub 2012 Jul 24. PMID 22829448
- [Result] Gletsu-Miller N, Kahn HS, Gasevic D, Liang Z, Frediani JK, Torres WE, Ziegler TR, Phillips LS, Lin E. Sagittal abdominal diameter and visceral adiposity: correlates of beta-cell function and dysglycemia in severely obese women. Obes Surg. 2013 Jul;23(7):874-81. doi: 10.1007/s11695-013-0874-6. PMID 23408092
- [Result] Phillips LS, Olson DE. Diabetes: normal glucose levels should be the goal. Nat Rev Endocrinol. 2012 Sep;8(9):510-2. doi: 10.1038/nrendo.2012.139. Epub 2012 Jul 31. No abstract available. PMID 22847240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Atlanta VA patients without known diabetes, who were at high risk of having unrecognized dysglycemia based on age >=45 years, BMI >=25 kg/m2, or other risk factors, were eligible for the study. Patients presenting for primary care visits were approached if they appeared to have age >=45 years and BMI >=25 kg/m2.
Groups:
- Group 1: Atlanta VA Medical Center patients who meet criteria for screening for prediabetes and early diabetes based on standard guidelines of the VA, American Diabetes Association, and NIH. This primarily included outpatient Veterans. Subjects were primarily included if they had age at least 45 years and BMI of 25 or greater, but some younger subjects were also included if they had risk factors for diabetes.
  Glucose challenge test: At a first outpatient visit, at different times of the day and without a prior fast, subjects will have a 50 gram glucose drink followed by measurement of plasma and capillary glucose along with A1c one hour later. They will also fill out questionnaires. At a second outpatient visit, in the morning after fasting overnight, they will have a 75 gram oral glucose tolerance test.
  Glucose tolerance test: Subjects found to have diabetes or prediabetes on the initial glucose tolerance test may be requested to have a repeat glucose tolerance test and A1c.
Period: Overall Study
Arm/Group | Group 1
Started | 1939
Consented | 1939 (consented)
Completed GCT Screening | 1876
Complete GCT, OGTT, A1c, Demographics | 1535
Completed | 1535
Not Completed | 404
Not completed — Failure to have the OGTT was most common | 404

BASELINE CHARACTERISTICS:
Population: Individuals receiving care at the Atlanta VA Medical Center
Groups:
- Group 1: Atlanta VA Medical Center patients who meet criteria for screening for prediabetes and early diabetes based on standard guidelines of the VA, American Diabetes Association, and NIH. This primarily included outpatient Veterans. Subjects were primarily included if they had age at least 45 years and BMI of 25 or greater, but some younger subjects were also included if they had risk factors for diabetes.
Arm/Group | Group 1
Number analyzed (Participants) | 1535
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 1441
Region of Enrollment [Number; unit: participants] — Individuals receiving care at the Atlanta VA Medical Center
  participants
    United States | 1535
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.3 (5.20)

OUTCOME MEASURES:

1. Primary Outcome: Ability of Different Screening Tests Which Can be Performed Opportunistically (During Outpatient Visits -- at Any Time of Day, Regardless of Meal Status) to Predict Findings With the Oral Glucose Tolerance Test (in the Morning, After an Overnight Fast)
Description: Area under ROC curve (AROC) for prediction of diabetes (based on OGTT) and high-risk dysglycemia (based on OGTT, IGT with 2 hour OGTT glucose 140-199 mg/dl, and/or IFG with fasting glucose 110-125 mg/dl).
  ROC curves are plots of (1-sensitivity) vs. (1-specificity) for all possible screening cutoffs, so a higher AROC indicates higher predictive accuracy. A perfect test would have an AROC of 1.00, while a test equivalent to tossing a coin (random) would have an AROC of 0.50; if confidence limits include 0.50, predictive accuracy is no better than chance.
  It is important to appreciate that while AROC analysis can show the relative accuracy of different screening tests, and aid the selection of which test to use in clinical practice, such an analysis does not define what the optimal screening test cutoff is. Selection of the optimal cutoff generally requires consideration of other factors, such as costs and/or the clinical importance of having higher or lower sensitivity.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: area under ROC curve
Groups:
- GCTpl - Diabetes; GCTpl - Dysglycemia: plasma glucose measured 1 hour after a 50g oral glucose challenge, performed at any time during the day, without requiring a prior overnight fast
- GCTcap - Diabetes; GCTcap - Dysglycemia: capillary glucose measured 1 hour after a 50g oral glucose challenge, performed at any time during the day, without requiring a prior overnight fast
- RPG - Diabetes: random plasma glucose measured prior to administration of the 50g oral glucose challenge, at any time during the day, without requiring a prior overnight fast
- RCG - Diabetes: random capillary glucose measured prior to administration of the 50g oral glucose challenge, at any time during the day, without requiring a prior overnight fast
- A1c - Diabetes; A1c - Dysglycemia: hemoglobin A1c, measured at the time of the OGTT
- RPG - Dysglycemia: random plasma glucose measured prior to the 50g oral glucose challenge, performed at any time during the day, without requiring a prior overnight fast
- RCG - Dysglycemia: random capillary glucose measured prior to the 50g oral glucose challenge, performed at any time during the day, without requiring a prior overnight fast
Arm/Group | GCTpl - Diabetes | GCTcap - Diabetes | RPG - Diabetes | RCG - Diabetes | A1c - Diabetes | GCTpl - Dysglycemia | GCTcap - Dysglycemia | RPG - Dysglycemia | RCG - Dysglycemia | A1c - Dysglycemia
Number analyzed (Participants) | 1535 | 1535 | 1535 | 1535 | 1535 | 1535 | 1535 | 1535 | 1535 | 1535
area under ROC curve | .85 [.78 to .91] | .82 [.75 to .89] | .76 [.69 to .82] | .72 [.65 to .80] | .67 [.57 to .76] | .76 [.72 to .80] | .73 [.69 to .77] | .66 [.62 to .71] | .64 [.59 to .68] | .63 [.58 to .68]

2. Secondary Outcome: Cost to Identify a Single Case of High-risk Dysglycemia or Previously Unrecognized Diabetes
Description: Cost was expressed as cost (dollars) to identify a single case, with cases defined as (i) diabetes or (ii) high-risk dysglycemia. Cost projections for screening were conducted from both Medicare and VA perspectives. All screening projections assumed follow-up testing with an OGTT if the screening test exceeded a 70% specificity cut-off.
Time Frame: 3 years
Measure: Number; unit: Dollars
Groups:
- GCTpl - Diabetes - VA: VA costs per case of diabetes identified, using the GCTpl screening test
- GCTcap - Diabetes - VA: VA costs per case of diabetes identified, using the GCTcap screening test
- GCTpl - Dysglycemia - VA: VA costs per case of dysglycemia identified, using the GCTpl screening test
- GCTcap - Dysglycemia - VA: VA costs per case of dysglycemia identified, using the GCTcap screening test
- GCTpl - Diabetes - Medicare: Medicare costs per case of diabetes identified, using the GCTpl screening test
- GCTcap - Diabetes - Medicare: Medicare costs per case of diabetes identified, using the GCTcap screening test
- GCTpl - Dysglycemia - Medicare: Medicare costs per case of dysglycemia identified, using the GCTpl screening test
- GCTcap - Dysglycemia - Medicare: Medicare costs per case of dysglycemia identified, using the GCTcap screening test
Arm/Group | GCTpl - Diabetes - VA | GCTcap - Diabetes - VA | GCTpl - Dysglycemia - VA | GCTcap - Dysglycemia - VA | GCTpl - Diabetes - Medicare | GCTcap - Diabetes - Medicare | GCTpl - Dysglycemia - Medicare | GCTcap - Dysglycemia - Medicare
Number analyzed (Participants) | 1535 | 1535 | 1535 | 1535 | 1535 | 1535 | 1535 | 1535
Dollars | 100 | 93 | 42 | 37 | 133 | 125 | 55 | 50

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/1939
Other Adverse Events (participants affected / at risk) | 11/1939
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=1939)
hypoglycemia during OGTT (Metabolism and nutrition disorders) | 7 (7) — glucose <50 mg/dl
hyperglycemia before 50g glucose challenge (Metabolism and nutrition disorders) | 2 (2) — capillary glucose >350 mg/dl
hyperglycemia after 50g glucose challenge (Metabolism and nutrition disorders) | 2 (2) — capillary glucose >350 mg/dl

LIMITATIONS AND CAVEATS:
Study in a single healthcare system, in a convenience sample of patients receiving care in a VA primary care clinic, in a population that was largely older, heavier, and predominantly male, and a single OGTT was used as the "gold standard".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes